CLINICAL TRIAL: NCT01907243
Title: The Role of Spreader Flaps in Preventing of Nasal Obstruction in Primary Rhinoplasty: A Randomized-controlled Trial.
Brief Title: The Role of Spreader Flaps in Preventing of Nasal Obstruction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Babak Saedi, Associate professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 91--02-48-6933
Record Dates: First submitted 2013-07-11; First posted 2013-07-24 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Nasal Obstruction
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- spreader flap (Active Comparator): Usage of spreader flap of upper lateral cartilage
  Interventions: Procedure: spreader flap
- Control group (No Intervention): performing of rhinoplasty without spreader flap

INTERVENTIONS:
Procedure: spreader flap — producing of upper lateral cartilage flap as a spreader flap
  Arms: spreader flap

SUMMARY:
Nasal obstruction is a preventable complication of rhinoplasty, for which the spreader graft is the gold standard. More recently, the spreader flap technique has been espoused as an alternative to spreader grafting. Herein we evaluated the efficacy of this technique in a randomized trial setting.

DETAILED DESCRIPTION:
Rhinoplasty is a common facial plastic surgery procedure, one complication of which is nasal vault narrowing and consequent nasal obstruction. Recently, researchers have paid much attention to nasal valve area and especially to the role of upper lateral cartilage (ULC) in preserving of nasal patency, since a possible consequence of destructive techniques was permanent functional problems for patients. In addition to functional problems, it can cause some aesthetic problems such as the inverted-V deformity . Accordingly, reconstruction of the midvault after dorsal reduction has been advocated and widely adopted.

The gold standard for midvault reconstruction after dorsal reduction has been the spreader graft, first advocated by Sheen . Subsequently, its usage has been widened to include repair of the valve in the unoperated nose, and its efficacy well-documented. However, it can be a time-consuming procedure that requires the harvest of septal cartilage. Therefore, some authors proposed the spreader flap as an alternative technique. While the results of the above mentioned articles proposed the efficacy of spreader flaps, none of them was a randomized trial and subjective methods were used for measurement of nasal breathing after rhinoplasty.

Nasal obstruction can be evaluated in different methods, both quantitative and subjective, the validity of each debated. For example, while the numeric form of Visual Analogue Scale (VAS) is commonly used, it is ultimately related to patients' subjective perception. Alternatively, objective evaluation of nasal patency is also of common interest to many researchers, and various methods for objective measurement exist. Among these different methods, acoustic rhinomanometry is an effective tool. However, some researchers debate the reliability of these results. Herein we examine the efficacy of the spreader flap in preventing nasal obstruction after dorsal reduction using a randomized trial with both objective and subjective measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent rhinoplasty

Exclusion Criteria:

* revision rhinoplasty
* congenital malformations
* severe allergic rhinitis
* nasal polyposis
* sinusitis
* deviated nose

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
acoustic rhinometry ( minimum cross section area) | before surgery
  acoustic rhinomanometery GM (ARI model, U.K) with an ultrasound system 0/8. (US-100, Japan) All tests were done while the patients were sitting while holding the device before his nose, completely sealing the nose, without excessive pressure cause changing of the nasal shape.
  Reducing the possible mucosal effect on acoustic rhinomanometry results, all tests were performed 10 minutes after the decongestant (Oxymetasoline spray) usage.
  Finally, a graph was drawn with two notches wherein the first notch related the valve area and the second one related to anterior part of lower turbinate. Each examination consisted of three consecutives tests from which the minimum cross section area was calculated

SECONDARY OUTCOMES:
acoustic rhinometry ( minimum cross section area) | one year after surgery
  coustic rhinomanometery GM (ARI model, U.K) with an ultrasound system 0/8. (US-100, Japan) All tests were done while the patients were sitting while holding the device before his nose, completely sealing the nose, without excessive pressure cause changing of the nasal shape.
  Reducing the possible mucosal effect on acoustic rhinomanometry results, all tests were performed 10 minutes after the decongestant (Oxymetasoline spray) usage.
  Finally, a graph was drawn with two notches wherein the first notch related the valve area and the second one related to anterior part of lower turbinate. Each examination consisted of three consecutives tests from which the minimum cross section area was calculated

CONTACTS AND LOCATIONS:
Overall Officials: Babak Saaedi, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Imam Khomeini Hospital, Tehran, Tehran Province, Iran